CLINICAL TRIAL: NCT03705325
Title: Evaluating Asthma Exacerbation-induced Changes in Lung Function With a Home-based Spirometer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VitalFlo Inc. (Industry)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VF-Cor2018
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Asthma; Asthma Attack; Asthma, Allergic
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: This is a prospective single arm study of 12-21 year olds with persistent asthma. Participants will be given the home spirometer and an iPhone 5S (without SIM card) loaded with the VitalFlo app. Participants will be asked to use the spirometer at least twice daily (in the morning between 6am and 10am and in the evening between 6am and 10pm) and whenever rescue medication (albuterol) is administered or the participant feels symptoms of asthma (such as cough, wheezing, or shortness of breath) in order to document lung function. After performing the spirometry maneuver, the user will be prompted to answer questions about their asthma symptoms. Changes in lung function will be matched to subject-reported asthma symptoms and/or albuterol use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Spirobank smart spirometer with VitalFlo mobile app (Experimental): In this single arm study, all participants will be receive the spirometer and an iPhone 5S (without SIM card) loaded with the VitalFlo app.
  Interventions: Device: Spirobank Smart spirometer

INTERVENTIONS:
Device: Spirobank Smart spirometer — The spirometer is a compact, portable, home-based spirometer that pairs with a smartphone app. Exhaled air flow causes the turbine to rotate, generating a voltage analogous to the rate of air flow across the turbine. The spirometer measures Forced expiratory volume in 1 second (FEV1), or the volume of air that is exhaled in the first second. The device prompts the user to perform a minimum of three expiratory maneuvers in and records the best of the three maneuvers. The information generated is then transmitted to the VitalFlo App (password protected) on the user's iPhone. The user is alerted, by the App, if their expiratory effort is inadequate (such as early termination of exhalation) and is provided coaching for proper technique.

SUMMARY:
The investigators will study the use of a home-based spirometer (Spirobank Smart spirometer) that connects to a smartphone app (VitalFlo) in teenagers with persistent asthma to determine if clinically significant changes in lung function detected by the spirometer are associated with patient-reported asthma symptoms.

DETAILED DESCRIPTION:
Asthma is a common chronic illness and significant expense to our healthcare system. Asthma affects nearly 25 million Americans, including 10% of U.S. adolescents. Teenagers are one of the most difficult groups to engage in self-management of chronic health problems like asthma and are at greater risk of poorly controlled asthma compared to younger children. Up to 80% of children with asthma are non-adherent to their controller medications, often due to lack of parent or child-perceived need or beneficial effects of these medications. Adolescents may have a higher threshold for initiating rescue treatment due to the perceived normalcy of asthma symptoms and frequently under-report symptoms to parents and healthcare providers.

Poor perception of asthma symptoms leads to overestimation of asthma control. Defining well controlled versus poorly controlled asthma is highly dependent on self-reported asthma symptoms. Up to half of patients with severe asthma symptoms report well controlled asthma. Many have low expectations of asthma control and have adapted to the disease so much so that they no longer perceive their limitations. Inaccurate self-reported data can be problematic in studies evaluating the impact of environmental factors or the efficacy of asthma treatments. An objective measure of asthma impairment is pulmonary function testing performed by spirometry. Ready access to a conventional spirometer is not always realistic in clinical care or research settings. The investigators propose integrating technology-based tools that leverage on the high rates of smartphone use among youth to identify early signs of deteriorating asthma control.

The Spirobank smart spirometer is a compact, portable, home-based spirometer approximately the size of an inhaler that pairs with a smartphone app called VitalFlo. The device uses an energy conserving turbine. Exhaled air flow causes the turbine to rotate, generating a voltage analogous to the rate of air flow across the turbine. The spirometer measures Forced expiratory volume in 1 second (FEV1), or the volume of air that is exhaled in the first second. The device prompts the user to perform a minimum of three expiratory maneuvers in and records the best of the three maneuvers. The information generated is collected on a microprocessor and then transmitted by a low power Bluetooth radio to the VitalFlo App (password protected) on the user's iPhone. The user is alerted, by the App, if their expiratory effort is inadequate (such as early termination of exhalation) and is provided coaching for proper technique. The data is then transmitted to a HIPAA-compliant cloud database. Participants will receive a survey after each time they measure lung function to gather information about any asthma symptoms they are experiencing. Investigators will ask that they use the spirometer prior to using albuterol for symptoms if possible. VitalFlo will also track, via cloud databases, outdoor temperature, humidity, air quality, and pollen counts: all environmental factors that can influence asthma symptoms. Routine calibration is not needed. The eventual goal of home spirometer use is to identify drops in lung function preceding asthma symptoms to allow persons with asthma to intervene with rescue medications early in hopes of preventing progression to a more serious exacerbation of asthma ("red zone") requiring healthcare utilization, such as emergency care or hospitalization.

This is a prospective single arm intervention study of 12-21 year olds with persistent asthma. Participants will be given the home spirometer after receiving instruction on proper use of the device. The participants will also receive an iPhone 5S (without SIM card) loaded with the VitalFlo app. Participants will be asked to use the spirometer at least twice daily (in the morning between 6am and 10am and in the evening between 6am and 10pm) and whenever rescue medication (albuterol) is administered or the participant feels symptoms of asthma (such as cough, wheezing, or shortness of breath) in order to document lung function. Pulmonary function testing is known to show diurnal variability. Investigators will use the morning and evening measurements to calculate the mean FEV1 for the day. After performing the spirometry maneuver, the user will be prompted to answer questions about their asthma symptoms. The lung function measurements and responses to the questions will be transmitted to a cloud-based HIPAA-compliant database and will be available for the investigators to download. Changes in lung function will be matched to subject-reported asthma symptoms and/or albuterol use.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 12 to 21 years, inclusive, of both genders
2. Physician diagnosis of persistent asthma or symptoms consistent with persistent asthma based on NHLBI Expert Panel Review 3 guidelines for diagnosis and management of asthma.
3. Current use of a controller therapy such as an inhaled corticosteroid (ICS), ICS in combination with long-acting beta agonist (LABA), or leukotriene receptor antagonist (LTRA).
4. A history of at least one asthma exacerbation requiring oral corticosteroids (OCS) in the past 12 months.
5. Wireless internet access in the participant's home

Exclusion Criteria:

1. Systemic corticosteroid-dependent asthma (i.e. people who take oral steroids such as prednisone daily for asthma control).
2. Pulmonary disease other than asthma that in the opinion of investigators may affect the interpretation of spirometry data, including but not limited to vocal cord dysfunction, restrictive lung disease, or cystic fibrosis.
3. Inability to perform spirometry.
4. History of spirometry-induced bronchoconstriction.
5. Pregnancy or nursing a baby.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-03 (Actual)

PRIMARY OUTCOMES:
change in FEV1 from baseline during "yellow zone" events | 6 months
  To determine if there is a clinically significant reduction from baseline in FEV1 percent predicted (for age, sex, height, and race) values obtained from the spirometer associated with "yellow zone" events, as defined by the participant's personalized asthma action plan. For the purposes of this study, we will define yellow zone events as any asthma symptoms (such as cough, wheezing, chest tightness) with or without use of rescue albuterol (excluding pre-exercise use of albuterol). A reduction of 10 percentage points or more in mean percent predicted FEV1 will be considered a clinically significant change.

SECONDARY OUTCOMES:
Correlation between change in FEV1 from baseline during yellow zone events and likelihood of experiencing unscheduled healthcare visits | 6 months
  To determine if the magnitude of the change from baseline in FEV1 associated with yellow zone events predicts unscheduled healthcare visits with the participant's primary care physician. Participants will be queried at each study visit about doctor's visits, emergency or urgent care visits, or hospitalizations related to asthma and whether or not oral steroids were prescribed

CONTACTS AND LOCATIONS:
Overall Officials: Allison Burbank, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - EPA Human Studies Facility, Chapel Hill, North Carolina
  - NC State Park Scholars Children's Specialty Clinic, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No